CLINICAL TRIAL: NCT04182139
Title: Acute Effects of Static Stretching Intensity and Duration on Muscle Viscoelastic Properties and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Yusuf Hasirci, Principal Investigator, Physiotherapist, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09.2018.479
Record Dates: First submitted 2019-08-18; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Static Stretching
Keywords: Static Stretching; Stiffness; Proprioception; Healthy adults
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 30 seconds and %50 intensity stretching (Experimental): The participants in this group performed an 30 seconds, %50 intensity static stretching exercise. 3 repetitive static stretching exercises did to hamstring muscles on the dominant side.
  Interventions: Other: Static Stretching Exercise
- 30 seconds and %75 intensity stretching (Experimental): The participants in this group performed an 30 seconds, %75 intensity static stretching exercise. 3 repetitive static stretching exercises did to hamstring muscles on the dominant side.
  Interventions: Other: Static Stretching Exercise
- 30 seconds and %100 intensity stretching (Experimental): The participants in this group performed an 30 seconds, %100 intensity static stretching exercise. 3 repetitive static stretching exercises did to hamstring muscles on the dominant side.
  Interventions: Other: Static Stretching Exercise
- 60 seconds and %50 intensity stretching (Experimental): The participants in this group performed an 60 seconds, %50 intensity static stretching exercise. 3 repetitive static stretching exercises did to hamstring muscles on the dominant side.
  Interventions: Other: Static Stretching Exercise
- 60 seconds and %75 intensity stretching (Experimental): The participants in this group performed an 60 seconds, %75 intensity static stretching exercise. 3 repetitive static stretching exercises did to hamstring muscles on the dominant side.
  Interventions: Other: Static Stretching Exercise
- 60 seconds and %100 intensity stretching (Experimental): The participants in this group performed an 60 seconds, %100 intensity static stretching exercise. 3 repetitive static stretching exercises did to hamstring muscles on the dominant side.
  Interventions: Other: Static Stretching Exercise

INTERVENTIONS:
Other: Static Stretching Exercise — Each intervention group received a different duration and intensity of static stretching exercise protocol.

SUMMARY:
The purpose of this study is to compare the acute effects of different duration and intensity of static stretching exercises on the viscoelastic properties of the hamstring muscle and the knee proprioception.

DETAILED DESCRIPTION:
Traditionally stretching exercises have been used by health professionals as a means of preventing injuries by increasing performance and increasing joint flexibility. Kubo et al. suggest that the potential mechanism of decreased risk of injury with increased flexibility is a change in the viscoelastic properties of the muscle-tendon unit. Muscle fibers and tendons contain proprioceptors. These receptors provide information about joint angle, muscle length and muscle tension. There are two stretch-related proprioceptors that transmit information to the central nervous system about muscle tension. These receptors are muscle spindles (respond to changes in the length) and golgi tendon organs (respond to changes in the tension). For this reason, interactions between muscle tension, muscle-tendon unit, viscoelasticity and proprioceptive tissue (muscle spindles and golgi tendon organ); it becomes important when you think about how stretching exercises affect proprioception, flexibility and increase or decrease of joint range of motion. In the literature, four stretching parameters have been defined as important to influence the potential for increasing or decreasing the flexibility of a joint: intensity, duration, frequency and stretching position. The focus of this study we plan on is the intensity and duration of stretching.

Exercise warming exercises before sportive activity and cooling exercises afterwards are widely suggested and applied. Determining the relationship between stretch severity and duration and viscoelastic properties and proprioception will contribute to the effective creation of training programs.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 18-45 age range.
* Volunteer to participate in the study.

Exclusion Criteria:

* Having had previous lower extremity operations.
* Having an orthopedic, neurological and rheumatologic disease of the lower extremities.
* Having open wound in the application area.
* Having had soft tissue injury in the last 6 weeks in the application area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline muscle viscoelastic properties at immediately after exercise | 10 minutes
  Muscle viscoelastic properties was assessed with Myoton® PRO device. It is an evidence-based device that evaluates the bio-mechanical properties of soft biological tissues in a non-invasive, objective, reliable, inexpensive, quick and easy manner. Myoton® PRO is used in studies to evaluate superficial skeletal muscles, connective tissues such as tendons and ligaments, and other soft tissues. It is a highly reliable method for assessing the tone, stiffness, elasticity of muscles.
Change from baseline proprioception at immediately after exercise | 10 minutes
  Proprioception was assessed with MarVAJED (Marmara Visual Auditory Joint Education Device). MarVAJED is a system for evaluating joint range of motion, analyzing joint position sense, offering biofeedback support to increase joint control, as well as directing it to controlled exercises. Analyzes joint movement with the help of small sensors. Transfers the obtained data to mobile phone, tablet or personal computer.
Change from baseline static stretching exercise intensity at the beginning of each exercise | 10 minutes
  A visual analog scale of 100 mm was used to assess the intensity of stretching exercise perceived by the participant at the beginning of each repetition. The visual analog scale is used to visually measure the intensity of the detected mechanical stimulus. 0 means "no stretch" and 100 means "maximum tolerable stretch without pain". Perceived violence from left to right increases.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Hasırcı, Principal Investigator — Marmara University; Semra Oğuz, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kubo K, Kanehisa H, Kawakami Y, Fukunaga T. Influence of static stretching on viscoelastic properties of human tendon structures in vivo. J Appl Physiol (1985). 2001 Feb;90(2):520-7. doi: 10.1152/jappl.2001.90.2.520. PMID 11160050
- [Background] Apostolopoulos N, Metsios GS, Flouris AD, Koutedakis Y, Wyon MA. The relevance of stretch intensity and position-a systematic review. Front Psychol. 2015 Aug 18;6:1128. doi: 10.3389/fpsyg.2015.01128. eCollection 2015. PMID 26347668